CLINICAL TRIAL: NCT07187661
Title: Efficacy of Intra-Articular Bevacizumab in Preventing Recurrent Hemarthrosis in Hemophilia Patients With Chronic Synovitis: A Pre- and Post-Design Study
Brief Title: Intra-Articular Bevacizumab for Preventing Recurrent Hemarthrosis in Hemophilia With Chronic Synovitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/006
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia; Chronic Synovitis
Keywords: Hemophilia A; Chronic Synovitis; Hemarthrosis; Hemophilic Arthropathy
MeSH Terms: conditions — Hemophilia A; Hemarthrosis | interventions — Bevacizumab; (18F)GTP1

STUDY DESIGN:
Intervention Model Description: This is an interventional clinical trial utilizing a pre- and post-study design. It is a single-arm study, meaning all enrolled participants will receive the investigational intervention. The trial is open-label, with no masking (blinding) of participants, care providers, investigators, or outcomes assessors. As it is a single-arm study, there is no allocation or randomization process. The total enrollment for this study is 25 participants.
Masking Description: This is an open-label study. No masking is used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-articular Bevacizumab (Experimental): All participants will receive intra-articular injections of Bevacizumab. The initial dose for the first four patients will be 20 mg/0.8 ml. If no major toxicities are observed, the dose will be escalated to 40 mg/1.6 ml for the remaining patients. Injections will be administered monthly for a duration of 4 months.
  Interventions: Drug: Intra-articular Bevacizumab

INTERVENTIONS:
Drug: Intra-articular Bevacizumab — This clinical trial investigates the intra-articular injection of Bevacizumab, a recombinant humanized monoclonal antibody that inhibits Vascular Endothelial Growth Factor (VEGF). The intervention functions by binding to and neutralizing VEGF-A, thereby blocking the pathogenic angiogenesis and vascular permeability that characterizes chronic hemophilic synovitis. For administration, the first four patients will receive a dose of 20 mg in 0.8 mL per injection, and if this is well-tolerated without major toxicities, the dose for all subsequent patients will be increased to 40 mg in 1.6 mL. Each injection will be administered directly into the target joint (knee, elbow, or ankle) once every 28 days for a total of four doses. Crucially, all injections will be performed only after appropriate prophylactic factor replacement to mitigate any procedure-related bleeding risk.
  Other Names: Avastin; Genentech

SUMMARY:
Hemophilia is an inherited bleeding disorder characterized by deficiency of clotting factors, leading to increased bleeding tendencies. The most common complications are joint bleeds (hemarthroses), which cause chronic changes in joints and ultimately disability. Recurrent hemarthroses often result from chronic synovitis in target joints of patients with hemophilia, a process driven by Vascular Endothelial Growth Factor (VEGF) mediated pathological angiogenesis. Intra-articular administration of Bevacizumab, a VEGF neutralizing monoclonal antibody, may block this process and reduce the frequency of recurrent joint bleeds. This study evaluates the efficacy and safety of intra-articular Bevacizumab for preventing recurrent hemarthrosis in patients with hemophilia and chronic synovitis.

DETAILED DESCRIPTION:
Hemophilia A is the most prevalent inherited bleeding disorder in Pakistan, accounting for approximately 69% of all hemophilia cases. A major complication is recurrent joint bleeding (hemarthrosis), which leads to chronic synovitis and progressive hemophilic arthropathy. This joint deterioration significantly impairs mobility and quality of life.

The underlying pathophysiology is driven by repeated hemarthroses, which cause increased local expression of Vascular Endothelial Growth Factor (VEGF). VEGF promotes abnormal angiogenesis and synovial proliferation, perpetuating a cycle of inflammation and bleeding, even when symptoms are not overt.

Bevacizumab is a recombinant humanized monoclonal antibody that specifically inhibits VEGF. Local intra-articular administration offers a targeted therapeutic approach to disrupt this pathogenic cycle directly at the site of pathology. By neutralizing VEGF, Bevacizumab may mitigate synovitis, reduce bleeding frequency, and slow progression of hemophilic arthropathy, while minimizing systemic exposure and associated adverse effects.

To investigate this therapeutic strategy, a two-year, open-label, single-arm clinical trial will be conducted at the Institute of Pathology and Diagnostic Medicine (IPDM), Khyber Medical University (KMU), and Hayatabad Medical Complex, Peshawar, Pakistan. A total of 25 participants with Hemophilia A and chronic synovitis in one or more target joints (knee, elbow, or ankle) will be enrolled.

All participants will receive intra-articular Bevacizumab injections following prophylactic factor replacement therapy to prevent procedure-related bleeding. The first four participants will receive 20 mg/0.8 mL per injection. If well tolerated without major toxicities, the remaining participants will receive 40 mg/1.6 mL per injection. Each injection will be administered into the target joint once every 28 days for a total of four doses.

The primary efficacy outcome will be the change in the Annualized Bleeding Rate (ABR) of the target joint, calculated from 3-month pre- and post-treatment data. Secondary outcomes will include changes in joint health assessed using the Hemophilia Joint Health Score (HJHS, Version 2.1; range 0-124, where higher scores indicate worse joint health) and synovial inflammation measured by Magnetic Resonance Imaging (MRI) with the International Prophylaxis Study Group (IPSG)-compatible scoring system.

This study may provide critical insight into a novel, VEGF-targeted strategy for managing chronic synovitis in hemophilia patients and preserving long-term joint health.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Hemophilia A.
* Presence of one or more target joints (knee, elbow, ankle) with chronic synovitis and a history of >2 hemarthrosis episodes in the past 6 months.
* Target joint World Federation of Hemophilia (WFH) joint score of 2-3.
* Adequate hematological, renal, and liver function (as specified by protocol lab values).
* Ability and willingness to provide informed consent and comply with the study protocol.

Exclusion Criteria:

* HIV positive diagnosis.
* Severely damaged joints or anatomical limitations preventing safe injection.
* Contraindications to MRI.
* Uncontrolled hypertension.
* Recent major surgery/trauma (<28 days).
* Serious non-healing wound, active cardiovascular disease, or other significant comorbidities that could increase risk or interfere with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) of the Target Joint | Baseline (3 months pre-treatment) compared to the 3-month period following the completion of the treatment protocol (i.e., 3 months after the 4th injection).
  The efficacy of the intervention will be assessed by the change in the number of recurrent hemarthrosis episodes specifically in the treated target joint. The rate will be annualized from data collected over a 3-month period. Response will be categorized as: 'Excellent' (0 bleeds), 'Good' (75-99% reduction), 'Fair' (50-74% reduction), or 'Poor' (<50% reduction).
Clinical Joint Health Score | Baseline scores compared to scores at 1, 3, 6, and 12 months after initiation of therapy
  Change in joint health and function as measured by the Hemophilia Joint Health Score (HJHS 2.1), a standardized physical examination tool that assesses pain, swelling, muscle atrophy, crepitus on motion, range of motion (flexion/extension loss), strength, and gait.
  Scale Range: 0 to 124 (higher scores indicate worse joint health and function).
  Interpretation:
  0 = best outcome (no joint damage or impairment)
  124 = worst outcome (severe joint involvement and functional limitation)
Synovial Hypertrophy | Baseline MRI (before starting therapy) compared to MRI performed 6 months after completion of therapy.
  Change in synovial membrane thickness in the target joint as assessed by MRI, scored according to the IPSG MRI scale for synovial hypertrophy (0-3; 0 = none, 3 = >5 mm).
Joint Effusion/Hemarthrosis | Baseline vs. 6 months after completion of therapy.
  Change in effusion or hemarthrosis volume in the target joint, assessed using the IPSG MRI scale (0-3; 0 = none, 3 = severe joint distention).
Synovial Inflammation Composite (Soft Tissue Subtotal) | Baseline vs. 6 months after completion of therapy.
  Change in the combined soft tissue inflammation score, calculated as the sum of effusion/hemarthrosis, synovial hypertrophy, and hemosiderin deposition (range 0-9)..

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kinza Ayaz, MBBS, Principal Investigator — Khyber Medical University Peshawar; Prof. Dr. Yasar M Yousafzai, PhD, Principal Investigator — Khyber Medical University Peshawar; Dr. Muhammad Tariq Masood Khan, MBBS, Principal Investigator — Khyber Medical University Peshawar; Dr Khalid Khan, MBBS, Principal Investigator — Khyber Medical University Peshawar
Locations (2):
- Pakistan (2):
  - Hayatabad Medical Complex, Peshawar, KPK
  - Institute of Pathology and Diagnostic Medicine (IPDM), Peshawar, KPK

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication (after de-identification) will be made available beginning 9 months following article publication and will remain available for a period of at least 36 months.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data will be made available 9 months after the publication of the primary results and will remain accessible for at least 36 months. Extensions may be considered upon request.
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Requestors will be required to submit a proposal to the corresponding author and sign a Data Access Agreement to ensure appropriate use of the data.

REFERENCES:
- [Background] Sadiq MA, Ahmed S, Afzal M, Tasfeen S. A basis for prenatal diagnosis of Haemophilia-A in Pakistani patients. Pak J Med Sci. 2022 Nov-Dec;38(8):2065-2070. doi: 10.12669/pjms.38.8.6524. PMID 36415265
- [Background] Hirayama AB, Silva AKCD, Rocha JS, Roberti MDRF. Prevalence of symptoms in hemophilia carriers in comparison with the general population: a systematic review. Hematol Transfus Cell Ther. 2019 Oct-Dec;41(4):349-355. doi: 10.1016/j.htct.2019.02.006. Epub 2019 Jun 17. PMID 31412987
- [Background] Gualtierotti R, Solimeno LP, Peyvandi F. Hemophilic arthropathy: Current knowledge and future perspectives. J Thromb Haemost. 2021 Sep;19(9):2112-2121. doi: 10.1111/jth.15444. Epub 2021 Jul 27. PMID 34197690
- [Background] Hassan S, Monahan RC, Mauser-Bunschoten EP, van Vulpen LFD, Eikenboom J, Beckers EAM, Hooimeijer L, Ypma PF, Nieuwenhuizen L, Coppens M, Schols SEM, Leebeek FWG, Smit C, Driessens MH, le Cessie S, van Balen EC, Rosendaal FR, van der Bom JG, Gouw SC. Mortality, life expectancy, and causes of death of persons with hemophilia in the Netherlands 2001-2018. J Thromb Haemost. 2021 Mar;19(3):645-653. doi: 10.1111/jth.15182. Epub 2020 Dec 18. PMID 33217158
- [Background] Iorio A, Stonebraker JS, Chambost H, Makris M, Coffin D, Herr C, Germini F; Data and Demographics Committee of the World Federation of Hemophilia. Establishing the Prevalence and Prevalence at Birth of Hemophilia in Males: A Meta-analytic Approach Using National Registries. Ann Intern Med. 2019 Oct 15;171(8):540-546. doi: 10.7326/M19-1208. Epub 2019 Sep 10. PMID 31499529